CLINICAL TRIAL: NCT05264272
Title: Disease Loads and Status of Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201904075RINA; 1103705906 (Dec23-2021 renew) (Other: National Taiwan University Hospital)
Record Dates: First submitted 2022-01-26; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Chronic Hepatitis B; Acute Hepatitis B; Hepatitis D
Keywords: hepatitis B; hepatitis D
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis D; Hepatitis B

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective Study: HBV/HDV positive individuals
  Interventions: Other: Prospective serological assays
- Retrospective Study: patients positive for anti-HDV
  Interventions: Other: Retrospective serological assays

INTERVENTIONS:
Other: Prospective serological assays — 1. Investigators will measure the levels of hemogram, AST, ALT, Bilirubine-total,Platelet, ALP, rGT, Albumin, GluAC, HBA1C, Albumin, INR, AFP, Creatinine, eGFR, HBsAg, quantitative HBsAg, anti-HBc, HBeAg, anti-HBe, HBV DNA, HBV genotype, anti-HDV, HDV RNA, and HDV RNA genotype at the enrollment of the study.
  2. BMI data, and Child-Pugh score (in cirrhotic patients) at the enrollment of the study. The smoking status, alcohol, coffee and green tea consumption, diabetes, family history of HCC will be collected.
  Groups: Prospective Study
Other: Retrospective serological assays — 1. Investigators will measure hemogram, AST, ALT, Bilirubine-total,Platelet, ALP, rGT, Albumin, GluAC, HBA1C, Albumin, INR, AFP, Creatinine, eGFR, HBsAg, quantitative HBsAg, anti-HBc, HBeAg, anti-HBe, HBV DNA, HBV genotype, anti-HDV, HDV RNA, HDV RNA genotype BMI data, and Child-Pugh score (in cirrhotic patients) at the enrollment of the study.
  2. The smoking status, alcohol, coffee and green tea consumption, diabetes, family history of HCC will be collected.
  Groups: Retrospective Study

SUMMARY:
The aim of study is to evaluate the current prevalence of HDV infection, and comprehensively analyze the interaction between HDV and HBV infections in the era of NAs in Taiwan. Investigators plan to set up a platform for HDV positive patients in Taiwan to invite sites or hepatologists who are interested in this field.

DETAILED DESCRIPTION:
Background The hepatitis Delta virus (HDV) was first discovered by Rizzetto at the end of the 1970s while a cohort of patients with hepatitis B virus (HBV) presented in Italy with severe hepatitis. HDV is a defective, single-stranded RNA virus, which required life-cycle function provided by the HBV. Therefore HDV infection can only occur in patients with HBV infection, either as simultaneous coinfection or superinfection. As compared with chronic HBV mono-infection, HBV and HDV dual infections leads to more severe liver disease, with increased rates of cirrhosis and hepatic decompensation, and an increased incidence of hepatocellular carcinoma (HCC).

It has been estimated that about 5% of chronic HBV carriers are coinfected by HDV, leading to an estimated 15-20 million people are HDV carriers worldwide. However, its prevalence varies in different geographic regions. Certain areas or countries have been described as high prevalence, such as Central and West Africa, Eastern Europe, the Middle East, Mongolia, Russia, and Vietnam. Taiwan is a high endemic country of HBV infection before the implementation of the universal infant hepatitis B immunization program, which was launched in 1984. Thereafter, the prevalence rate of HBV infection decreased from 20% to 12% in the population with age more than 35 years. After 30-year of national HBV vaccination program, the prevalence of HDV infection in general population remains low, from 5-8% in 1986 to 4.4% in 2012. However, there was a significant decrease in the incidence of acute HDV superinfection in the general population, from 23.7% in 1983 to 4.2% in 1995. It is worth noting that the significant increased prevalence of HDV infection among injection drug users (IDUs), particular in those with human immune-deficiency virus (HIV) infection.

Currently treatment options of HDV infection remain limited, and interferon remains in standstill as the only available treatment. Relapse could still be observed after the treatment. Combination of nucleos(t)ide analogues (NAs) with IFN did not provide any benefit compared with IFN mono-therapy. Currently there are three novel therapeutic approaches for chronic HDV infection, namely Myrcludex B, lonafarnib, and REP2139-Ca. Of them, the REP 2139 in combination with PegIFN induced the clearance of serum HDV-RNA and of HBsAg in about half of the patients, followed by the raising of anti-HBs. If the preliminary data are confirmed, the combination of Peg IFN with REP 2139 will represent in the therapy of CHD in the near future. Therefore, an updated prevalence of HDV infection, especially in high endemic country of HBV infection, is needed to further understand the condition of CHD in Taiwan.

Patients and Methods I. Part 1 Prospective Study Investigators will organize a multicenter, prospective study platform to enroll all the HBV/HDV positive individuals from referral hepatology centers in Taiwan. A blood sample will be drawn at the time of the visit, after getting the approval of IRB. After centrifugation, the serum will be stored at -80°C, and sent for HDV RNA test. The PIs will review all HBsAg-positive individuals before the enrollment of this study. Demographics, clinical and laboratory data and the patient's history will be collected in a common database. Diagnosis of cirrhosis is based on the liver biopsy（Metavir F4 or Ishak ≧ 5）or liver ultrasonographic evidence of cirrhosis with signs of portal hypertension (splenomegaly or presence of esophageal or gastric varices) or fibroscan >12kPa. The diagnosis of HCC is based on the criteria of practice guidelines of the European Association for the Study of the Liver (EASL) or the American Association for the Study of Liver Disease (AASLD). The fibroscan will be performed in patients with anti-HDV seropositivity.

Laboratory Test

1. Investigators will measure the levels of hemogram, AST, ALT, Bilirubine-total,Platelet, ALP, rGT, Albumin, GluAC, HBA1C, Albumin, INR, AFP, Creatinine, eGFR, HBsAg, quantitative HBsAg, anti-HBc, HBeAg, anti-HBe, HBV DNA, HBV genotype, anti-HDV, HDV RNA, and HDV RNA genotype at the enrollment of the study.
2. BMI data, and Child-Pugh score (in cirrhotic patients) at the enrollment of the study. The smoking status, alcohol, coffee and green tea consumption, diabetes, family history of HCC will be collected.
3. Investigators will collect 10cc serum. Serology The presence of HBsAg, HBeAg, anti-HCV antibodies, and anti-HDV antibodies will be determined using commercial assay kits (HBsAg EIA, Abbott, North Chicago, IL; HBeAg EIA, Abbott; anti-HCV, EIA 3.0, Abbott; anti-HDV, ELISA, GBC). HBsAg titers will be quantified with ElecsysHBsAg II Quant reagent kits (Roche Diagnostics, Indianapolis, IN) according to the manufacturer's instructions with a lower limit of detection of 0.05 IU/ml. HBV DNA will be quantified using the COBAS TaqMan HBV test (CAP-CTM; Roche Molecular Systems, Inc., Branchburg, NJ, USA) with a lower limit of detection of 20 IU/ml. Serum HDV RNA will be detected using in-house PCR, as previously described, with a lower limit of detection 400 copies/mL.

HBV and HDV genotyping HBV genotypes will be determined using restriction fragment length polymorphism on the surface gene of HBV (between nucleotide positions 256 and 796), as previously described. HDV genotypes will also be determined by using the PCR-restriction fragment length polymorphism method, as described previously.

HDV RNA II. Part 2 Retrospective Study Investigators will collect clinical data for patients positive for anti-HDV from Sep.2018~Dec.2019. Investigators will collect the following data if available in the chart :levels of hemogram, AST, ALT, Bilirubine-total,Platelet, ALP, rGT, Albumin, GluAC, HBA1C, Albumin, INR, AFP, Creatinine, eGFR, HBsAg, quantitative HBsAg, anti-HBc, HBeAg, anti-HBe, HBV DNA, HBV genotype, anti-HDV, HDV RNA, and HDV RNA genotype at the enrollment of the study.

BMI data, and Child-Pugh score (in cirrhotic patients) at the enrollment of the study. The smoking status, alcohol, coffee and green tea consumption, diabetes, family history of HCC will be collected.

Statistical analyses Statistical tests used in this study are Student t test and the chi-square square test. In addition, multivariate analysis will be used for estimating the odds ratios (ORs) and 95% confidence intervals (CIs). All of these tests are two sided, and the significance levels are set at a P value < 0.05. All statistical analysis will be performed using the SPsS statistical package (SPSS Inc., Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Chronic HBV
* Acute HBV
* anti-HDV positive

Exclusion Criteria:

* Other diagnostics deemed not suitable for this study by the principal investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hepatitis B and hepatitis D patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
HDV infection prevalence | 36 months
  The aim of study is to evaluate the current prevalence of HDV infection, and comprehensively analyze the interaction between HDV and HBV infections in the era of NAs in Taiwan.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No